CLINICAL TRIAL: NCT04129749
Title: Influence of Fatigue on the Walking Pattern in Cerebral Palsy Patients.
Status: Withdrawn | Type: Observational
Why Stopped: cancelled study
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Other Study IDs: 19-HPNCL-01
Record Dates: First submitted 2019-04-04; First posted 2019-10-17 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Real-Time Analysis Interactive Lab: walk spontaneously or at prescribed speeds of cerebral palsy patient to a standstill in a virtual and secure virtual reality environment.
  Interventions: Procedure: Real-Time Analysis Interactive Lab

INTERVENTIONS:
Procedure: Real-Time Analysis Interactive Lab — The Real-Time Analysis Interactive Lab uses an instrumented treadmill, a motion capture system (Vicon System), an electromyographic system as well as a virtual environment is projected on a 180 ° screen. This equipment allows patients to walk spontaneously or at prescribed speeds to a standstill in a virtual and secure virtual reality environment.

SUMMARY:
To date, studies do not study the influence of external disturbing factors on the market.

The main hypothesis is that the stopping of walking in paralyzed cerebral patients is mainly due to an increase in the energy cost of walking.

The secondary objectives are to study the causes of the increase in the energy cost of walking (modification of muscle coordination / increase of co-activations, loss of strength, etc.).

This study will use the GRAIL combining an instrumented treadmill, a motion capture system (Vicon System), an electromyographic system as well as a virtual environment projected on a 180 ° screen

DETAILED DESCRIPTION:
In most studies, the study of the gait of cerebral palsy patients is done through quantified walking analysis tests, objectively evaluating the kinetic and kinematic parameters, associated with the measurement of respiratory exchanges and heart rate.

Nevertheless this very objective evaluation does not really reflect the child's ability to perform the acts of everyday life that he wishes, and in particular, his ability to walk a long time.

It therefore appears that patients do not only want to walk better on an objective and analytical level but also aim to walk longer and improve their walking efficiency.

To date, studies do not study the influence of external disturbing factors on the market.

The main hypothesis is that the stopping of walking in paralyzed cerebral patients is mainly due to an increase in the energy cost of walking.

The main objective is to confirm this hypothesis. The secondary objectives are to study the causes of the increase in the energy cost of walking (modification of muscle coordination / increase of co-activations, loss of strength, etc.).

For that, the investigators will use a tool that is perfectly adapted: the GRAIL (Real-Time Analysis Interactive Lab). The GRAIL uses an instrumented treadmill, a motion capture system (Vicon System), an electromyographic system as well as a virtual environment is projected on a 180 ° screen. This equipment allows patients to walk spontaneously or at prescribed speeds to a standstill in a virtual and secure virtual reality environment. Throughout the duration of the test, the investigators will quantify the evolution of biomechanical (kinematic, kinetic and EMG) and physiological (gas analysis system) factors during walking.

This is a study conducted in a usual evaluation framework: market analysis is commonly indicated for paralyzed children, in order to assess their disability and to propose the best therapy. There was no inherent risk in the proposed study protocol, but possible fatigue is inevitably analyzed, which is not related to inclusion in this study.

ELIGIBILITY:
Inclusion Criteria:

* children aged 7 to 18 years (diplegic, hemiparetic or tetraparetic) requiring treatment with botulinum toxin
* followed at the Lenval Foundation
* walking alone more than 6 minutes
* parental information and no disagreement

Exclusion Criteria:

* Modification of spasticity treatments within 6 months of evaluation: baclofen pump, oral baclofen, retraction surgery (tenotomy, tendon lengthening, arthrodesis ...)
* dyskinesia
* Cognitive disorders in children that do not allow the use of GRAIL
* Contraindication to Botulinum Toxin (myasthenia, hypersensitivity and infections)
* Contraindication to physical activity (intercurrent pathology)

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: cerebral palsy patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-11-17 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Measure of energy cost during walk in cerebral palsy patients, by evolution of inter-segmental angle | at baseline Day 0
  Measure of energy cost during walk in cerebral palsy patients by quantify modification of muscle coordination / increase of co-activations, loss of strength of muscle.
  This will be evaluated by the evolution of inter-segmental angles (degrees) during a 6 minutes walking test.
Measure of energy cost during walk in cerebral palsy patients, by evolution of articular force | at baseline Day 0
  Measure of energy cost during walk in cerebral palsy patients by quantify modification of muscle coordination / increase of co-activations, loss of strength of muscle.
  Also evaluated by the evolution of articular force (N/kg) during a 6 minutes walking test.
Measure of energy cost during walk in cerebral palsy patients by evolution of articular moment | at baseline Day 0
  Measure of energy cost during walk in cerebral palsy patients by quantify modification of muscle coordination / increase of co-activations, loss of strength of muscle.
  Also evaluated by the evolution of articular moment (N.m/kg) during a 6 minutes walking test.
Measure of energy cost during walk in cerebral palsy patients by evolution of articular power | at baseline Day 0
  Measure of energy cost during walk in cerebral palsy patients by quantify modification of muscle coordination / increase of co-activations, loss of strength of muscle.
  Also evaluated by the evolution of articular power (W/kg) during a 6 minutes walking test

SECONDARY OUTCOMES:
quantification of biomechanical factors during walking by evolution of inter-segmental angles | at baseline Day 0
  Measure of kinematic and kinetic parameters during walk in cerebral palsy patients.
  This will be evaluated by the evolution of inter-segmental angles (degrees) during a 6 minutes walking test.
quantification of biomechanical factors during walking by evolution of articular force | at baseline Day 0
  Measure of kinematic and kinetic parameters during walk in cerebral palsy patients.
  This will be evaluated by the evolution of articular force (N/kg) during a 6 minutes walking test.
quantification of biomechanical factors during walking by evolution of articular moment | at baseline Day 0
  Measure of kinematic and kinetic parameters during walk in cerebral palsy patients.
  This will be evaluated by the evolution of articular moment (N.m/kg) during a 6 minutes walking test.
quantification of biomechanical factors during walking by evolution of of articular power | at baseline Day 0
  Measure of kinematic and kinetic parameters during walk in cerebral palsy patients.
  This will be evaluated by the evolution of of articular power (W/kg) during a 6 minutes walking test.
measure of physiological factors during walking by evolution of oxygen consummation | at baseline Day 0
  measure of O2 consummation during walk in cerebral palsy patients by a gas system analysis.
  This will be evaluated by the evolution of O2 consummation during walk during a 6 minutes walking test.
measure of physiological factors during walking by evolution of carbon dioxide consummation | at baseline Day 0
  measure of CO2 consummation during walk in cerebral palsy patients by a gas system analysis.
  This will be evaluated by the evolution of CO2 consummation during walk during a 6 minutes walking test..

CONTACTS AND LOCATIONS:
Overall Officials: RAMPAL Virginie, MD, Principal Investigator — Fondation Lenval - Nice Children Hôpitaux Pédiatriques de Nice
Locations (1):
- Hôpitaux Pédiatriques de Nice CHU-Lenval, Nice, France